CLINICAL TRIAL: NCT00976573
Title: A Randomized Phase II Trial of Carboplatin, Paclitaxel, Bevacizumab, With or Without Everolimus for Therapy of Metastatic Malignant Melanoma
Brief Title: Carboplatin, Paclitaxel, and Bevacizumab With or Without Everolimus in Treating Patients With Metastatic Malignant Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N0879; NCI-2011-01968 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000654465 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Results first posted 2017-03-07 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Melanoma (Skin)
Keywords: Stage IV Skin Melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — Bevacizumab; Carboplatin; Everolimus; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (bevacizumab, paclitaxel, and carboplatin) (Experimental): Patients receive bevacizumab IV over 30-90 minutes on days 1 and 15, paclitaxel IV over 60 minutes on days 1, 8, and 15, and carboplatin IV over 30 minutes on day 1. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: bevacizumab; Drug: carboplatin; Drug: paclitaxel
- Arm II(bevacizumab, paclitaxel, carboplatin, and everolimus) (Experimental): Patients receive bevacizumab, paclitaxel, and carboplatin as in Arm I. Patients also receive everolimus PO QD on 3 days a week. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: bevacizumab; Drug: carboplatin; Drug: everolimus; Drug: paclitaxel

INTERVENTIONS:
Biological: bevacizumab — Given IV
Drug: carboplatin — Given IV
Drug: everolimus — Given orally
  Arms: Arm II(bevacizumab, paclitaxel, carboplatin, and everolimus)
Drug: paclitaxel — Given IV

SUMMARY:
This randomized phase II trial is studying how well carboplatin, paclitaxel, and bevacizumab work when given with or without everolimus in treating patients with malignant melanoma that has spread from where it started to other places in the body. Drugs used in chemotherapy, such as carboplatin and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, may block the ability of tumor cells to grow and spread. Everolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. It is not yet known whether combination chemotherapy given together with bevacizumab is more effective with or without everolimus in treating patients with metastatic melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess whether there is sufficient promise of an impact of the addition of everolimus to the combination of carboplatin, paclitaxel, and bevacizumab on progression-free survival that it would be recommended for further testing in patients with metastatic malignant melanoma.

Secondary

* To estimate the confirmed tumor response rate of each of the treatment regimens.
* To estimate the distribution of overall survival (OS) time for each of the treatment regimens.
* To assess the impact on the safety profile of the addition of everolimus to the combination of carboplatin, paclitaxel, and bevacizumab.

OUTLINE: This is a multicenter study. Patients are stratified according to elevated LDH (above upper limit of normal) at baseline (yes vs no), location of metastatic disease (M1a [skin, subcutaneous tissue, or lymph node only] vs M1b [lung] vs M1c [other visceral sites]) and prior chemotherapy for metastatic disease (yes vs no). Patients are randomized to 1 of 2 treatment arms.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive bevacizumab intravenously (IV) over 30-90 minutes on days 1 and 15, paclitaxel IV over 60 minutes on days 1, 8, and 15, and carboplatin IV over 30 minutes on day 1. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive bevacizumab, paclitaxel, and carboplatin as in Arm I. Patients also receive everolimus orally (PO) once daily (QD) 3 times weekly. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3-6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologic proof of stage IV malignant melanoma not amenable to surgery; (biopsy can be of locoregional disease in setting of clinically evident stage IV disease, but primary tumor alone will not qualify)
* At most one prior chemotherapy based regimen for metastatic melanoma (no prior taxane-based regimens allowed); note: prior adjuvant non-taxane based chemotherapy and/or adjuvant immunotherapy are allowed; no limit on the number of prior biologic, immunologic or targeted therapies
* Measurable disease defined as at least one lesion whose longest diameter can be accurately measured as >= 2.0 cm with chest x-ray, or as >= 1.0 cm with computed tomography (CT) scan, CT component of a positron emission tomography (PET)/CT, or magnetic resonance imaging (MRI) scan; note: disease that is measurable by physical examination only is not eligible
* Life expectancy >= 4 months
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Absolute neutrophil count (ANC) >= 1500/mL
* Platelets (PLT) >= 100,000 x 10^9/L
* Hemoglobin (Hgb) >= 9 g/dL (patients may be transfused to meet this requirement)
* Total cholesterol =< 300 mg/dL and; (note: serum levels of cholesterol or triglycerides found to be elevated may be lowered with anti-lipid therapy, but must be documented to be below these levels prior to enrollment)
* Triglycerides =< 2.5 X upper limit of normal (ULN); (note: serum levels of cholesterol or triglycerides found to be elevated may be lowered with anti-lipid therapy, but must be documented to be below these levels prior to enrollment)
* Creatinine =< 1.5 x ULN
* Total bilirubin =< 1.5 mg/dL (exception: patients with documented Gilbert's syndrome are allowed to participate despite elevated bilirubin)
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) =< 2.5 x ULN
* Alkaline phosphatase =< 2.5 x ULN
* Urine protein:creatinine (UPC) ratio < 1.0 at screening OR
* Urine dipstick for proteinuria < 2+ (patients discovered to have >= 2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate =< 1 g of protein in 24 hours to be eligible)
* Negative pregnancy test done =< 7 days prior to registration/randomization, for women of childbearing potential only
* Ability to understand and the willingness to sign a written informed consent document
* Willing to return to a North Central Cancer Treatment Group (NCCTG) institution for follow-up
* Willing to provide mandatory blood samples for research purposes
* Willing to follow a diet low in fat and cholesterol while taking everolimus
* Willing to abstain from eating grapefruit or drinking grapefruit juice for the duration of the study

Exclusion Criteria

* Prior treatment with agents disrupting vascular endothelial growth factor (VEGF) activity (i.e., bevacizumab, VEGF-trap, anti-VEGF receptor [R] monoclonal antibody [Mab]) or targeting VEGFR (e.g. sunitinib, sorafenib)
* Prior treatment with an mTOR inhibitor for melanoma (sirolimus, temsirolimus, everolimus)
* Brain metastases per MRI or CT at any time prior to registration; note: patients that have had primary therapy for brain metastasis (i.e. surgical resection, whole brain radiation, or stereotactic radiation therapy [SRT] even if stable) are not eligible
* Other investigational agents =< 4 weeks prior to registration/randomization
* Chemotherapy treatment =< 3 weeks prior to registration/randomization
* Any biologic, immunologic or targeted therapy =< 2 weeks prior to registration/randomization
* Major surgical procedure, open biopsy, or significant traumatic injury =< 4 weeks prior to registration/randomization
* Fine needle aspirations or core biopsies =< 7 days prior to registration/randomization
* Planned/or anticipated major surgical procedure during the course of the study
* Other medical conditions including but not limited to:

  * History of liver disease such as cirrhosis, chronic active hepatitis, chronic persistent hepatitis or hepatitis B or C
  * Active infection requiring parenteral antibiotics
  * Poorly controlled high blood pressure (>=150 mm Hg systolic and/or 100 mmHg diastolic) despite treatment
  * New York Heart Association class II-IV congestive heart failure
  * Serious cardiac arrhythmia requiring medication
  * Myocardial infarction or unstable angina =< 6 months prior to registration/randomization
  * Clinically significant peripheral vascular disease
  * Deep venous thrombosis or pulmonary embolus =< 1 year of registration/randomization and/or ongoing need for full-dose oral or parenteral anticoagulation
  * Ongoing anti-platelet treatment other than low-dose aspirin (i.e., aspirin 81 mg orally [p.o.] daily)
  * Active bleeding or pathological conditions that carry high risk of bleeding (e.g., known esophageal varices, etc.)
  * Serious, non-healing wound (including wounds healing by secondary intention), ulcer or bone fracture
  * History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess =< 6 months prior to registration/randomization
  * History of central nervous system (CNS) disease (e.g., primary brain tumor, vascular abnormalities, etc.), clinically significant stroke or transient ischemic attack (TIA) =< 6 months prior to registration/randomization, seizures not controlled with standard medical therapy
  * Radiographically documented tumor invading major blood vessels
  * History of hypertensive crisis or hypertensive encephalopathy
  * Uncontrolled diabetes as defined by fasting serum glucose > 1.5 x ULN
  * Severely impaired lung function as defined as spirometry and diffusing capacity of the lung for carbon monoxide (DLCO) that is 50% of the normal predicted value and/or 02 saturation that is 88% or less at rest on room air
  * A known history of human immunodeficiency virus (HIV) seropositivity
* Any of the following as this regimen may be harmful to a developing fetus or nursing child:

  * Pregnant women
  * Nursing women
  * Men and women of reproductive potential who are not using effective birth control methods must use highly effective contraception throughout the trail and for 6 months after last study treatment
* Existence of peripheral sensory neuropathy >= grade 2
* History of other malignancy =< 5 years with the exception of basal cell or squamous cell carcinoma of the skin, treated with local resection only, or carcinoma in situ (e.g. of the cervix, breast, prostate, etc.)
* =< 4 weeks since last day of adjuvant radiation therapy prior to registration or =< 2 weeks since last day of palliative radiation therapy; NOTE: patients who have had > 25% of their functional bone marrow irradiated are not eligible for this trial
* Active or recent history of hemoptysis (>= 1/2 teaspoon of bright red blood per episode) =< 30 days prior to registration
* Known hypersensitivity to any of the components of the everolimus, bevacizumab, carboplatin, or paclitaxel
* Current use of drugs that are known to be strong inhibitors or inducers of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4); note: if these agents are discontinued, everolimus therapy can begin >= 7 days after discontinuation of such agent
* Positive hepatitis B antigen (HBsAg) or hepatitis C serology (HCV) tests
* Planned immunization with attenuated live vaccines =< 7 days prior to registration or during study period; note: close contact with those who have received attenuated live vaccines should be avoided during treatment with everolimus; examples of live vaccines include intranasal influenza, measles, mumps, rubella, oral polio, Bacillus Calmette-Guérin (BCG), yellow fever, varicella and TY21a typhoid vaccines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2010-04; Primary Completion 2014-12 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert McWilliams, MD, Study Chair — Mayo Clinic
Locations (310):
- United States (310):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Contra Costa Regional Medical Center, Martinez, California
  - El Camino Hospital Cancer Center, Mountain View, California
  - Bay Area Breast Surgeons, Incorporated, Oakland, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Larry G Strieff MD Medical Corporation, Oakland, California
  - Tom K Lee, Incorporated, Oakland, California
  - Doctors Medical Center - San Pablo Campus, San Pablo, California
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Michael and Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - Lakeland Regional Cancer Center at Lakeland Regional Medical Center, Lakeland, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - John B. Amos Cancer Center, Columbus, Georgia
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Illinois CancerCare - Bloomington, Bloomington, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare - Canton, Canton, Illinois
  - Illinois CancerCare - Carthage, Carthage, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Illinois CancerCare - Eureka, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Illinois CancerCare - Havana, Havana, Illinois
  - Illinois CancerCare - Kewanee Clinic, Kewanee, Illinois
  - La Grange Memorial Hospital, La Grange, Illinois
  - Illinois CancerCare - Macomb, Macomb, Illinois
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - Moline, Illinois
  - Illinois CancerCare - Monmouth, Monmouth, Illinois
  - OSF Holy Family Medical Center, Monmouth, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Illinois CancerCare - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Illinois CancerCare - Pekin, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare - Peru, Peru, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Illinois CancerCare - Princeton, Princeton, Illinois
  - Illinois CancerCare - Spring Valley, Spring Valley, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Elkhart Clinic, LLC, Elkhart, Indiana
  - Michiana Hematology-Oncology, PC - Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - St. Francis Hospital Cancer Care Services, Indianapolis, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Michiana Hematology-Oncology, PC - South Bend, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center, Mishawaka, Indiana
  - Michiana Hematology Oncology PC - Plymouth, Plymouth, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC - La Porte, Westville, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Bettendorf, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, Clive, Iowa
  - Mercy Cancer Center - West Lakes, Clive, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's Hospital - South, Overland Park, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - CCOP - Kansas City, Prairie Village, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Boston University Cancer Research Center, Boston, Massachusetts
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - Mercy General Health Partners, Muskegon, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Lakeside Cancer Specialists, PLLC, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - MeritCare Bemidji, Bemidji, Minnesota
  - St. Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Duluth Clinic, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology - Woodbury, Woodbury, Minnesota
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Goldschmidt Cancer Center, Jefferson City, Missouri
  - Saint Luke's Cancer Institute at Saint Luke's Hospital, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology Oncology Associates, Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Mercy Clinic Cancer and Hematology - Rolla, Rolla, Missouri
  - Saint Joseph Oncology, Incorporated, Saint Joseph, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Charles R. Wood Cancer Center at Glens Falls Hospital, Glens Falls, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Moses Cone Regional Cancer Center at Wesley Long Community Hospital, Greensboro, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - FirstHealth Moore Regional Community Hospital Comprehensive Cancer Center, Pinehurst, North Carolina
  - Annie Penn Cancer Center, Reidsville, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Wood County Oncology Center, Bowling Green, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Community Cancer Center, Elyria, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Southern Ohio Medical Center Cancer Center, Portsmouth, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Cancer Care Associates - Norman, Norman, Oklahoma
  - Cancer Care Associates - Mercy Campus, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Geisinger Hazleton Cancer Center, Hazleton, Pennsylvania
  - Guthrie Cancer Center at Guthrie Clinic Sayre, Sayre, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Cancer Centers of the Carolinas - Faris Road, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Grove Commons, Greenville, South Carolina
  - Greenville Hospital Cancer Center, Greenville, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Greer Medical Oncology, Greer, South Carolina
  - Cancer Centers of the Carolinas - Seneca, Seneca, South Carolina
  - Cancer Centers of the Carolinas - Spartanburg, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Danville Regional Medical Center, Danville, Virginia
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Mary Babb Randolph Cancer Center at West Virginia University Hospitals, Morgantown, West Virginia
  - Center for Cancer Treatment & Prevention at Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Care at Regional Cancer Center, Eau Claire, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Saint Joseph's Hospital, Marshfield, Wisconsin
  - Marshfield Clinic - Lakeland Center, Minocqua, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Ministry Medical Group at Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - St. Nicholas Hospital, Sheboygan, Wisconsin
  - Marshfield Clinic at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Saint Michael's Hospital Cancer Center, Stevens Point, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin

REFERENCES:
- [Derived] Slostad JA, Liu MC, Allred JB, Erickson LA, Rumilla KM, Block MS, Keppen M, King D, Markovic SN, McWilliams RR. BRAF V600 Mutation Detection in Plasma Cell-Free DNA: NCCTG N0879 (Alliance). Mayo Clin Proc Innov Qual Outcomes. 2021 Oct 13;5(6):1012-1020. doi: 10.1016/j.mayocpiqo.2021.05.003. eCollection 2021 Dec. PMID 34703985

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A (Bevacizumab, Paclitaxel, and Carboplatin): Patients receive 10 mg/kg bevacizumab IV over 30-90 minutes on days 1 and 15, 80 mg/m^2 paclitaxel IV over 60 minutes on days 1, 8, and 15, and AUC 5 carboplatin IV over 30 minutes on day 1. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Arm B (Bevacizumab, Paclitaxel, Carboplatin, and Everolimus): Patients receive bevacizumab, paclitaxel, and carboplatin as in Arm I. Patients also receive 5 mg everolimus PO QD three times weekly (e.g. Monday, Wednesday, Friday). Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Arm A (Bevacizumab, Paclitaxel, and Carboplatin) | Arm B (Bevacizumab, Paclitaxel, Carboplatin, and Everolimus)
Started | 75 | 74
Completed | 71 | 71
Not Completed | 4 | 3
Not completed — Ineligible | 0 | 1
Not completed — Cancel prior to receiving treatment | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Bevacizumab, Paclitaxel, and Carboplatin) | Arm B (Bevacizumab, Paclitaxel, Carboplatin, and Everolimus) | Total
Number analyzed (Participants) | 75 | 74 | 149
Age, Continuous [Median (Full Range); unit: years] | 59 [26 to 85] | 58 [29 to 81] | 59 [26 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 33 | 54
  Male | 54 | 41 | 95
Region of Enrollment [Number; unit: participants]
  United States | 75 | 74 | 149

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: The primary endpoint is progression-free survival (PFS) defined as the time from randomization to documentation of disease progression or death without documentation of progression. The distribution of PFS times will be estimated using the Kaplan-Meier method. Progression is defined using the RECIST Criteria as at least a 20% increase in the sum of diameters of target lesions taking as reference the smallest sum of diameters recorded on study (this includes the baseline sum if that is the smallest on study) or the appearance of one or more new lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm of target lesions, or the appearance of one or more new lesions, unequivocal progression of existing non-target lesions, although unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.
Time Frame: Time from randomization to documentation of disease progression or death without documentation of progression;Up to 5 years
Population: Intent-to-treat analysis population: All participants enrolled are included in the primary analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Bevacizumab, Paclitaxel, and Carboplatin) | Arm B (Bevacizumab, Paclitaxel, Carboplatin, and Everolimus)
Number analyzed (Participants) | 75 | 74
months | 5.6 [4.7 to 8.3] | 5.1 [3.9 to 6.7]

2. Secondary Outcome: Toxicity
Description: For this secondary endpoint, toxicity is defined as a grade 3 or higher adverse events that is classified as either possibly, probably, or definitely related to study treatment. The assignment of attribution to study treatment and grade (or degree of severity) of the adverse event are classified using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. The percentage of participants reporting a grade 3 or higher toxicity is reported. For a list of all reported adverse events, please refer to the Adverse Events Section below.
Time Frame: Up to 5 years
Population: Participants who completed the study (specified in the Participant Flow) are included.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A (Bevacizumab, Paclitaxel, and Carboplatin) | Arm B (Bevacizumab, Paclitaxel, Carboplatin, and Everolimus)
Number analyzed (Participants) | 71 | 71
percentage of participants
  Neutropenia | 35 | 58
  Leukopenia | 17 | 24
  Fatigue | 11 | 17

3. Secondary Outcome: Confirmed Tumor Response Rate (Complete Response [CR] or Partial Response [PR]) According to Response Evaluation Criteria in Solid Tumors (RECIST) Criteria
Description: Confirmed Tumor Response: A confirmed tumor response is defined to be a CR or PR (by the RECIST criteria) noted as the objective status on 2 consecutive evaluations at least 8 weeks apart. The proportion of tumor responses will be estimated by the number of confirmed tumor responses divided by the total number of evaluable patients. A ninety percent confidence interval for the true proportion of confirmed tumor responses will be calculated assuming that the number of confirmed tumor responses follows a binomial distribution.
Time Frame: Up to 5 years
Population: Intent-to-treat analysis population: All participants enrolled are included.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm A (Bevacizumab, Paclitaxel, and Carboplatin) | Arm B (Bevacizumab, Paclitaxel, Carboplatin, and Everolimus)
Number analyzed (Participants) | 75 | 74
percentage of patients | 13 [6.0 to 22.7] | 23 [13.5 to 34.0]

4. Secondary Outcome: Overall Survival Time
Description: Overall survival time is defined as the time from registration to death due to any cause. The distribution of survival times will be estimated using the method of Kaplan-Meier.
Time Frame: up to 5 years
Population: Intent-to-treat analysis population: All participants enrolled are included.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Bevacizumab, Paclitaxel, and Carboplatin) | Arm B (Bevacizumab, Paclitaxel, Carboplatin, and Everolimus)
Number analyzed (Participants) | 75 | 74
months | 14.5 [11.5 to 21.8] | 10.8 [9.1 to 14.3]

ADVERSE EVENTS:
Time Frame: Adverse events are assessed less than or equal to 14 days prior to registration, prior to each cycle of treatment, at discontinuation of study treatment, and during observation 28-42 days after discontinuation of study treatment; Up to 5 years.
Description: The CTEP Version 4.0 of the NCI Common Terminology Criteria for Adverse Events (CTCAE) will be utilized for AE reporting. All graded adverse events are reported. Patients who completed the study (as specified in the Participant Flow) and had adverse events assessed are included below.
Arm/Group | Arm A (Bevacizumab, Paclitaxel, and Carboplatin) | Arm B (Bevacizumab, Paclitaxel, Carboplatin, and Everolimus)
Serious Adverse Events (participants affected / at risk) | 12/71 | 18/71
Other Adverse Events (participants affected / at risk) | 71/71 | 71/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Bevacizumab, Paclitaxel, and Carboplatin) (N=71) | Arm B (Bevacizumab, Paclitaxel, Carboplatin, and Everolimus) (N=71)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Jejunal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (2) | 1 (1)
Death NOS (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
Flu like symptoms (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1)
Anaphylaxis (Immune system disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 4 (4) | 5 (5)
Platelet count decreased (Investigations) | 2 (2) | 2 (2)
White blood cell decreased (Investigations) | 2 (2) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (3) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 1 (2)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Lymphedema (Vascular disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Bevacizumab, Paclitaxel, and Carboplatin) (N=71) | Arm B (Bevacizumab, Paclitaxel, Carboplatin, and Everolimus) (N=71)
Anemia (Blood and lymphatic system disorders) | 63 (357) | 59 (332)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 1 (1) | 2 (2)
Dry eye (Eye disorders) | 1 (1) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 24 (51) | 24 (47)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 9 (11) | 5 (7)
Diarrhea (Gastrointestinal disorders) | 7 (12) | 10 (16)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 2 (6)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 2 (3)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 3 (11) | 8 (11)
Nausea (Gastrointestinal disorders) | 40 (152) | 46 (129)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 22 (46) | 25 (52)
Death NOS (General disorders) | 1 (1) | 1 (1)
Edema limbs (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 68 (408) | 67 (352)
Fever (General disorders) | 14 (19) | 15 (16)
Infusion related reaction (General disorders) | 2 (7) | 0 (0)
Infusion site extravasation (General disorders) | 0 (0) | 2 (2)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 10 (14) | 7 (8)
Anaphylaxis (Immune system disorders) | 0 (0) | 1 (1)
Anorectal infection (Infections and infestations) | 0 (0) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 2 (3) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 1 (1)
Lip infection (Infections and infestations) | 1 (1) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Peripheral nerve infection (Infections and infestations) | 0 (0) | 1 (1)
Rash pustular (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 3 (3)
Sinusitis (Infections and infestations) | 1 (3) | 2 (6)
Skin infection (Infections and infestations) | 2 (2) | 5 (7)
Soft tissue infection (Infections and infestations) | 1 (2) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (3) | 3 (4)
Urinary tract infection (Infections and infestations) | 1 (3) | 2 (2)
Vulval infection (Infections and infestations) | 0 (0) | 1 (2)
Wound infection (Infections and infestations) | 2 (2) | 1 (1)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (4) | 3 (9)
Alanine aminotransferase increased (Investigations) | 0 (0) | 3 (3)
Alkaline phosphatase increased (Investigations) | 0 (0) | 3 (4)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 3 (3)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
CD4 lymphocytes decreased (Investigations) | 2 (2) | 1 (2)
Cholesterol high (Investigations) | 0 (0) | 6 (13)
Creatinine increased (Investigations) | 2 (3) | 2 (2)
Investigations - Other, specify (Investigations) | 1 (2) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 5 (14) | 7 (13)
Lymphocyte count increased (Investigations) | 1 (1) | 1 (1)
Neutrophil count decreased (Investigations) | 49 (177) | 59 (209)
Platelet count decreased (Investigations) | 47 (177) | 50 (196)
Weight gain (Investigations) | 1 (12) | 2 (2)
Weight loss (Investigations) | 2 (3) | 5 (23)
White blood cell decreased (Investigations) | 54 (217) | 55 (215)
Anorexia (Metabolism and nutrition disorders) | 8 (14) | 13 (23)
Dehydration (Metabolism and nutrition disorders) | 7 (8) | 4 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1) | 11 (34)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 6 (6)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 3 (7)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 4 (7) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (5) | 2 (11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 (41) | 24 (60)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (6)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 14 (28) | 25 (66)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (6) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2)
Dysesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 3 (7) | 7 (12)
Headache (Nervous system disorders) | 1 (3) | 3 (3)
Hypersomnia (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Olfactory nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (9) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 2 (2) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 36 (190) | 29 (159)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (4) | 2 (6)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 14 (24) | 14 (31)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Irregular menstruation (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (28) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 13 (32) | 21 (73)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Nail loss (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (4) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 39 (190) | 37 (205)
Hypotension (Vascular disorders) | 1 (1) | 5 (5)
Peripheral ischemia (Vascular disorders) | 1 (2) | 0 (0)
Thromboembolic event (Vascular disorders) | 4 (5) | 5 (9)
Vascular disorders - Other, specify (Vascular disorders) | 0 (0) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes